CLINICAL TRIAL: NCT03852082
Title: Predictors and Clinical Outcomes of Patients With Coronary Heart Disease Co-morbid Depression Post Percutaneous Coronary Intervention
Acronym: PCICODE
Status: Active, not recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Vice President, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: 20180317
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Coronary Heart Disease; Percutaneous Coronary Intervention; Depression
MeSH Terms: conditions — Coronary Disease; Depression | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: percutaneous coronary intervention — Patients with coronary heart disease co-morbid depression post percutaneous coronary intervention.

SUMMARY:
A prospective, multicenter, registered cohort study to observe the incidence of 1-year major adverse cardiac events in patients with coronary heart disease co-morbid depression treated with percutaneous coronary intervention and to clarify the predictors of 1-year major adverse cardiac events post PCI among these patients.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is a clinical relevant psychosomatic issue. Treatment strategies include percutaneous coronary intervention (PCI), guidelines medication (GDMT) and coronary artery bypass grafting (CABG) were clinical proven to be effective to realize myocardial revascularization post CHD. Previous studies revealed that diagnosed depressed CHD patients have 3.6 times higher risk of major adverse events (MACE) post percutaneous coronary intervention than nondepressed. However, a reliable explanation of how depression impact clinical outcomes of CHD patients post PCI is lacking. The objective of this study is to observe the incidence of major adverse cardiovascular events in patients with coronary heart disease co-morbid with depression post PCI, and to explore a prognostic model of clinical outcomes based on physiological, interventional, socio-economic and psychological factors among these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures;
2. Men and women 18 years or older；
3. Diagnosed CHD needed to and can be treated with PCI according to the guidelines of ACC/AHA；
4. Willingness to participate in the follow-up study for at least 1 year.

Exclusion Criteria:

1. Inability to provide written informed consent;
2. Diagnosed mental illness or medical history (including schizophrenia, bipolar disorder, severe dementia or Lifetime alcohol or substance abuse);
3. Tendency of suicide;
4. Pregnant or lactating women;
5. Any physical or intellectual inability or disability that may affect completion of self-assessment tools, study protocol and follow-up requirements;
6. Any other reasons that investigators based on professional judgments that would place the patient at increased risk.
7. Patient with STEMI within 24-hour from the onset of chest pain to admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary heart disease co-morbid depression post percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2019-08-28 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Major Adverse Events | 36-month
  major adverse events were including all-cause mortality, myocardial infarction, in-stent thrombosis and target vessel revascularization.

SECONDARY OUTCOMES:
Number of Participants with All-cause Mortality | 36-month
Number of Participants with Cardiovascular Mortality | 36-month
Number of Participants with Myocardial Infarction | 36-month
Number of Participants with In-Stent Thrombosis | 36-month
Number of Participants with Target-Lesion Revascularization | 36-month

CONTACTS AND LOCATIONS:
Overall Officials: Shaoliang Chen, phd, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No